CLINICAL TRIAL: NCT05688254
Title: Internet-Based Stress Recovery Program for Adolescents
Acronym: FOREST-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (1.5 E) 250000-S-646
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-01

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated either to the intervention or control groups. The intervention group will use the intervention and the control will take care as usual.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will get a 4-week online stress recovery intervention.
  Interventions: Behavioral: FOREST-A
- Control group (No Intervention): The control group will take care as usual.

INTERVENTIONS:
Behavioral: FOREST-A — The internet-based psychosocial intervention will be delivered. The intervention comprises six modules: introduction, relaxation, psychological detachment, mastery, control, and summary, within psychoeducation and exercises in each module. The interactions with psychologists will be on demand. The whole intervention duration will be 4 weeks.
  Arms: Intervention group

SUMMARY:
The study aims to evaluate the feasibility and efficacy of the internet-based stress recovery program for adolescents.

DETAILED DESCRIPTION:
The FOREST-A is a third-wave cognitive behavioral therapy and mindfulness-based internet-delivered 4-week psychosocial intervention for recovery from stress, which was initially developed for healthcare workers and is now adapted for adolescents. The program comprises six modules: introduction, relaxation, psychological detachment, mastery, control, and summary, with psychologist engagement on-demand. Each module includes psychoeducation and exercises. The program will be delivered in Lithuanian.

The intervention will be evaluated using the two-arm randomized controlled trial with intervention and care as usual condition at pre-test and post-test.

ELIGIBILITY:
Inclusion Criteria:

* Recent exposure to life-stressor.
* Students of high schools in Lithuania.
* Comprehending Lithuanian.
* Parental and own consent for minor-aged participants (< 18 years)/only own consent for adolescents aged 18 years or older to participate in the study provided.
* Have access to a device (such as a tablet, phone or computer) with an internet connection.

Exclusion Criteria:

* Acute psychiatric condition/crisis.
* No recent life-stressor exposure, or low levels of stress.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The Recovery Experience Questionnaire | Pre-treatment, post-treatment (after 4 weeks), 3 months follow-up
  The Recovery Experience Questionnaire (Sonnentag & Fritz, 2007) adapted Child and Adolescent version will be used to measure the changes in recovery from stress experience. It is a self-report measure comprising 16 items, with provided 5-point Likert scale, ranging from Totally disagree (=1) to Totally agree (=5). Total scores may range from 16 to 80, and higher scores will indicate higher recovery.

SECONDARY OUTCOMES:
The Adjustment Disorder New Module-8 Child and Adolescent Version Questionnaire | Pre-treatment, post-treatment (after 4 weeks), 3 months follow-up
  The Adjustment Disorder New Module-8 Child and Adolescent Version (Kazlauskas et al., 2018) will be used to measure the changes in symptoms of adjustment disorder, which are described in the International Classification of diseases 11th edition (WHO, 2018). The measure includes a list of 16 potentially stressful events (with binary answers Yes and No, indicating whether the participant has experienced a stressor) and 8 items for adjustment disorder symptoms evaluation (with a 4-point Likert scale ranging from Never (=1) to Often (=4)). Total scores may range from 8 to 32, and higher scores will indicate higher adjustment problems.
The Generalized Anxiety Disorder-7 scale | Pre-treatment, post-treatment (after 4 weeks), 3 months follow-up
  The Generalized Anxiety Disorder-7 scale (Spitzer, Kroenke, Williams, & Löwe, 2007) will be used to measure the changes in generalized anxiety symptoms.The measure comprises 7 items with the possible answers ranging on a 4-point Likert scale from Not at all (=0) to Nearly every day (=3). Total scores may range from 0 to 21. Higher scores will indicate higher generalized anxiety symptoms.
The Patient Health Questionnaire-9 questionnaire | Pre-treatment, post-treatment (after 4 weeks), 3 months follow-up
  The Patient Health Questionnaire-9 (Löwe, Kroenke, Herzog, & Gräfe, 2004) will be used to measure changes in depressive symptoms. The measure comprises 9 items, with provided a 4-point Likert scale, ranging from Not at all (=0) to Nearly every day (=3). Total scores may range from 0 to 27. Higher scores will indicate higher depressive symptoms.
The WHO-5 Well-being Index Questionnaire | Pre-treatment, post-treatment (after 4 weeks), 3 months follow-up
  The WHO-5 Well-being Index (Topp, Østergaard, Søndergaard, & Bech, 2015) will be used to measure changes in general psychological well-being. The measure comprises 5 items with a Likert scale ranging At no time (=0) to All of the time (=5). Total scores may range from 0 to 25. Higher scores will indicate better psychological well-being.
The Perceived Positive Social Support Scale | Pre-treatment, post-treatment (after 4 weeks), 3 months follow-up
  The Perceived Positive Social Support Scale (Kazlauskas et al., 2022) will be used to measure changes in social support. The measure comprises 4 items, with provided an 8-point Likert scale ranging from Never (=0) to Always (=7). Total scores may range from 0 to 28. Higher scores will indicate higher perceived positive support.

OTHER OUTCOMES:
Program evaluation questions | Post-treatment (after 4 weeks)
  Participants will be given questions regarding the usage, general satisfaction, usefulness of the program, and subjective impact on psychological and physical well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Zelviene, PhD, Principal Investigator — Vilnius University, Institute of Psychology
Locations (1):
- Vilnius University, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zelviene P, Kairyte A, Dumarkaite A, Nomeikaite A, Kazlauskas E. Internet-based stress recovery intervention for adolescents: study protocol for a randomized controlled trial. Trials. 2023 Mar 8;24(1):174. doi: 10.1186/s13063-023-07188-1. PMID 36890560